CLINICAL TRIAL: NCT07235098
Title: Effect of a Music Intervention in Reducing Distress and Pain in Patients With Suspected or Diagnosed Lung Cancer Undergoing Mini-Invasive Surgery
Brief Title: Effect of a Music Intervention in Reducing Distress and Pain in Patients With Lung Cancer Undergoing Mini-invasive Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IOSI-MUSICAL-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Suspected or Confirmed)
Keywords: lung cancer; pain; anxiety; music
MeSH Terms: conditions — Lung Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a monocentric open-label randomized controlled clinical trial with two arms:
  * Arm A: classical music therapy + standard of care (SOC)
  * Arm B: SOC only Patients scheduled for minimally invasive lung resection, with a suspected or confirmed diagnosis of lung cancer, will be enrolled and randomized to one of the two arms of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A treated with classical music therapy and standard of care (Experimental): Patients with suspected or diagnosed lung cancer undergoing minimally invasive lung resection will be treated with classical music therapy and standard of care.
  Interventions: Other: Music therapy intervention
- Arm B treated with standard of care only (No Intervention): Patients with suspected or diagnosed lung cancer undergoing minimally invasive lung resection will be treated with standard of care only.

INTERVENTIONS:
Other: Music therapy intervention — Patient randomized to experimental Arm A will receive a classical music therapy intervention throughout the duration of their hospital stay for a minimally invasive lung resection.
  Arms: Arm A treated with classical music therapy and standard of care

SUMMARY:
This study aims at evaluating whether music therapy intervention is effective in decreasing psychological (distress) and physical symptoms (pain) in patients with suspected or diagnosed lung cancer undergoing minimally invasive lung surgery.

DETAILED DESCRIPTION:
A diagnosis of cancer may result in extensive emotional, physical and social suffering. Moreover, surgical treatment of lung cancer represents itself a stressful event. It is important that cancer care incorporates services that help meet patients' psychological, social and spiritual needs. Music therapy interventions have been used to alleviate symptoms and treatment side effects in cancer patients and their efficacy has been demonstrated in various settings. Within the distinction between music therapy (a personalized approach based on the interaction with a trained music therapist) and music medicine (with pre-recorded music), the best efficacy results have been reported with music therapy.

The use of music listening is growing in the field of music therapy intervention because of the impact musical contents can have on physiological, psychological and behavioural levels.

The primary objective of this study is to evaluate whether music therapy intervention is effective in decreasing psychological (distress) and physical symptoms (pain) in patients with suspected or diagnosed lung cancer undergoing minimally invasive lung surgery. Secondary objectives are the evaluation of the decrease of the serum cortisol as biomarker of stress and the request of additional doses of analgesics for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed diagnosis of lung cancer
* Age ≥ 18 years
* Indication for lung resection through a minimally invasive surgery
* Signed written informed consent

Exclusion Criteria:

* Endocrinological disorders involving cortisol axis
* Chronic steroid intake > 10 mg/day
* Concomitant treatment with drugs against symptomatic anxiety and/or depression
* Partial or complete hearing loss
* Inability to follow the schedule of investigation
* Patient unwilling to refrain from actively listening to other music (e.g., via other personal devices/headphones) outside of the prescribed musical intervention defined by the study protocol during the hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of distress | From the day of surgery until the day of discharge from the hospital (in average 6 days after surgery)
  Change of the level of distress on the Distress thermometer
Pain intensity | From the day of surgery until the day of discharge from the hospital (in average 6 days after surgery)
  Change of pain intensity on the numerical scale

SECONDARY OUTCOMES:
Serum cortisol levels | From the day of surgery until the day of discharge from the hospital (in average 6 days after surgery)
  Change in the levels of serum cortisol measured in the morning
Additional doses of analgesics for pain control | From the day of surgery until the day of discharge from the hospital (in average 6 days after surgery)
  Number of additional doses of analgesics administered for pain control per day

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided